CLINICAL TRIAL: NCT00225706
Title: Efficacy and Safety Study of Caldolor in Hospitalized Febrile Pediatric Patients
Brief Title: A Study of Caldolor in Hospitalized Febrile Pediatric Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cumberland Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPI-CL-005
Record Dates: First submitted 2005-09-22; First posted 2005-09-26 (Estimated); Last update posted 2010-04-12 (Estimated); Status verified 2007-10

CONDITIONS: Fever
MeSH Terms: conditions — Fever | interventions — Ibuprofen

INTERVENTIONS:
Drug: Caldolor

SUMMARY:
The primary objective of this study of Caldolor administered to febrile hospitalized pediatric patients every 6 hours for 24 hours is to determine the clinical equivalence of a single dose of Caldolor compared to acetaminophen (paracetamol; APAP) for the treatment of fever as measured by the AUC Tº within the first 6 hours of treatment (as compared to a target temperature of 98.6ºF [37.0ºC]).

ELIGIBILITY:
Inclusion Criteria:

1. Be hospitalized
2. Be between 6 months and 17 years of age, inclusive
3. Have new (not chronic, within last 7 days) onset of fever, documented by temperature greater than or equal to 101.0ºF (38.3ºC) (The preferred method of temperature measurement is core. The route of temperature measurement used immediately before randomization should be used immediately before dosing and for all temperature measurements during the Treatment Period.)
4. Have written informed consent provided by legal parent, guardian, or authorized agent, and have same agree to abide by the study restrictions and to return for the required assessments (Where appropriate, participants of appropriate intellectual maturity should personally provide written informed assent; age of assent may be determined by Institutional Review Boards (IRBs) or Independent Ethics Committees (IECs) or be consistent with local legal requirements.)

Exclusion Criteria:

1. Have inadequate intravenous access
2. Have received antipyretic drug therapy within 8 hours before dosing
3. Be pregnant or nursing
4. Have any history of allergy or hypersensitivity to NSAIDs, aspirin, APAP, or any component of Caldolor or APAP.
5. Have a history of severe head trauma that required the current hospitalization, had intracranial surgery or stroke within the previous 30 days, or have any history of intracerebral arteriovenous malformation, cerebral aneurysm, or central nervous system mass lesions
6. Have a history of febrile convulsion or have a sibling with a history of febrile convulsion
7. Have a history of congenital bleeding diatheses (e.g., hemophilia) or any active clinically significant bleeding, or have underlying platelet dysfunction, including (but not limited to) idiopathic thrombocytopenic purpura, disseminated intravascular coagulation, or congenital platelet dysfunction
8. Have gastrointestinal bleeding that has required medical intervention within the previous 6 weeks, unless definitive surgery has been performed
9. Have platelet count less than 30,000/mm3
10. Be receiving full dose anticoagulation therapy (Prophylaxis with subcutaneous heparin is acceptable.)
11. Have fever secondary to blood or drug reaction
12. Have an expected life span of less than 14 days because of imminent withdrawal of life support or severity of illness
13. Be receiving ongoing or imminent treatment with corticosteroids
14. Have neurogenic fever
15. Be on dialysis, have oliguria or calculated creatinine clearance of less than 70 mL/min (calculated using the Schwartz formula), have impaired renal function, be receiving nephrotoxic drugs, or be expected to be unable to tolerate the extra fluid required for administration of CTM
16. Have had major surgery within the past 12 hours, unless adequate hemostasis has been achieved
17. Have received another investigational drug within the past 30 days
18. Be otherwise unsuitable for the study, in the opinion of the Investigator

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2005-10; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Temperature

CONTACTS AND LOCATIONS:
Locations (3):
- Vanderbilt University Children's Hospital, Nashville, Tennessee, United States
- Hospital Cecilio Castillero, Chitré, Herrera Province, Panama
- Unitas Hospital, Lyttleton, Pretoria, South Africa